CLINICAL TRIAL: NCT06207123
Title: A Phase I/II Study to Investigate the Combination of LP-118, Ponatinib, Vincristine and Dexamethasone in Relapsed/Refractory T-ALL/LBL
Brief Title: A Study to Investigate LP-118, Ponatinib, Vincristine and Dexamethasone in Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma (LBL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-1382
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Acute Leukemia; Lymphoblastic Leukemia; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib; Vincristine; Dexamethasone; Calcium Dobesilate; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Participants (Single Arm) (Experimental): All study participants will receive LP-118 and ponatinib. The initial dose of LP-118 to be tested is 100 mg, and initial dose of ponatinib to be tested is 30 mg. Higher doses of LP-118 will only be tested if the study doctor feels it is safe to do so. A member of the study team will let study participants know which doses they are assigned.
  Study drugs will be given in 21-day cycles. There will be 7 study visits in cycle 1 (on Days 1, 5, 6, 7, 15, 22, and 28). LP-118 and ponatinib will be taken at home every day. Dexamethasone will be taken between days 1-7 and days 15-22. For Cycles 2-12, study participants will have 5 study visits per cycle (on Days 1, 8, 15, 22, and 28). On all days, study participants will take LP-118 and ponatinib at home.
  Participants in this group will also receive standard of care vincristine, dexamethasone, and methotrexate during study cycles.
  Interventions: Drug: LP-118; Drug: Ponatinib; Drug: Vincristine; Drug: Dexamethasone; Drug: Methotrexate

INTERVENTIONS:
Drug: LP-118 — LP-118 is an experimental anti-cancer drug that is currently being studied in clinical trials for multiple types of hematological cancers and solid tumors.
Drug: Ponatinib — Ponatinib is used to treat certain types of chronic myeloid leukemia (CML; a type of cancer of the white blood cells).
  Other Names: Iclusig
Drug: Vincristine — Vincristine is a chemotherapy medication used to treat various types of cancer, including leukemia, lymphoma, neuroblastoma, and Wilms tumor. Vincristine belongs to the category of vinca alkaloids, a class of drugs that function by impeding the proper division of cancer cells.
  Other Names: Oncovin; Vincrex; Vincasar PES
Drug: Dexamethasone — Dexamethasone is used to treat cancer, to decrease inflammation and sometimes used before and after chemotherapy to prevent or treat nausea and/or vomiting. It is given in the vein (IV) or orally (by mouth)
  Other Names: DexPak; Decadron
Drug: Methotrexate — Methotrexate is a drug used to treat cancer of the blood, bone, lung, breast, head, and neck. It can also treat rheumatoid arthritis and psoriasis.
  Other Names: Otrexup; Xatmep; Rasuvo

SUMMARY:
The purpose of this study is to learn more about LP-118 (an experimental drug) and its side effects and decide on acceptable doses. The purpose of this study is to determine if LP-118 can be given safely with another medicine called ponatinib, that is FDA-approved for the treatment of acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about LP-118 (an experimental drug) and its side effects and decide on acceptable doses. The purpose of this study is to determine if LP-118 can be given safely with another medicine called ponatinib, that is FDA-approved for the treatment of acute lymphoblastic leukemia.

This study will investigate the combination of LP-118 and ponatinib at different dose levels to find the best doses that can be safely given to patients. This means that enrolled subjects will receive progressive increasing or decreasing doses of these drugs until the maximally tolerated dose is determined. All participants will also receive a standard of care chemotherapy combination consisting of the FDA approved drugs vincristine, dexamethasone and intrathecal (injection into the spinal canal, also called "spinal tap") methotrexate. This combination is standard of care for relapsed T-ALL/LBL.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory patients with T-lineage acute lymphoblastic leukemia or T-lymphoblastic lymphoma
2. 18 years old or older
3. Bone marrow or peripheral blood involvement with ≥5% lymphoblasts or measurable residual disease with >10-4 level detected by multiparameter flow cytometry or next-generation sequencing (NGS)-based measurable residual disease (ClonoSEQ, Adaptive Technologies). Patients with isolated extramedullary disease that is measurable by computed tomography (CT) scan are also eligible.
4. Eastern Cooperative Oncology Group performance status 0-2.
5. Adequate organ function as defined by all of the following:

   1. Creatinine clearance ≥50 mL/min, determined by the Cockroft-Gault formula, or measured by a 24-hour urine collection.
   2. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN) and bilirubin ≤1.5 x ULN (unless considered due to Gilbert's syndrome or of non-hepatic origin i.e,, leukemic involvement). For patients with Gilbert's syndrome, bilirubin ≤1.5 x of their baseline bilirubin level will be required.
6. Participants must be at least 2 weeks from major surgery or radiation therapy. A wash-out period of 4 half-lives is required for patients who participated in other investigational trials. These patients must have recovered from clinically significant toxicities related to these prior treatments.
7. Participants must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.
8. Females of childbearing potential will use effective contraception during protocol treatment and for at least 8 months after the last dose. Males with female partners of reproductive potential will use effective contraception during protocol treatment and for at least 5 months after the last dose. A patient is of childbearing potential if, in the opinion of the treating investigator, he/she is biologically capable of having children and is sexually active. Female patients who are not of childbearing potential (ie, meet at least one of the following criteria):

   a. Have undergone hysterectomy or bilateral oophorectomy; or have medically confirmed ovarian failure; or are medically confirmed to be post-menopausal (cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause).
9. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Active central nervous system (CNS) leukemia
2. Active or chronic hepatitis B or C infection as evidenced by hepatitis B surface antigen and anti-hepatitis C antibody positivity, respectively, or known seropositivity for human immunodeficiency virus (HIV). Patients with HIV but an undetectable viral load are eligible for enrollment.
3. Major surgery within <2 weeks before randomization.
4. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function or unstable pulmonary condition.
5. Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix, or localized prostate cancer that has been definitely treated with radiation or surgery. Patients with previous malignancies are eligible provided that they have been disease free for ≥2 years or are not currently requiring treatment.
6. Uncontrolled cardiac disease.
7. Pregnant females; breastfeeding females; males with female partners of reproductive potential and females of childbearing potential not using highly effective contraception or not agreeing to continue highly effective contraception for a minimum of 5 months after the last dose of investigational product if male and 8 months after the last dose of investigational product if female.
8. Participation in other investigational studies during active treatment phase.
9. Other severe acute, chronic medical, psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the treating physician, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose To demonstrate safety and to identify the recommended phase II dose for combination of LP-118, ponatinib, vincristine and dexamethasone | 36 weeks
  Recommended phase II dose for combination of LP-118, ponatinib, vincristine and dexamethasone as assessed by rate of dose-limiting toxicities among study participants.

SECONDARY OUTCOMES:
Complete Clinical Remission at Days 28 and 56 | 36 weeks
  Complete clinical remission at days 28 and 56 for study participants defined as the disappearance of leukemia as indicated by <5% marrow blasts and the absence of peripheral blasts, with recovery of hematopoiesis defined by ANC ≥1000/μL and platelets ≥100,000/μL.
Complete clinical remission with incomplete count recovery (CRi) at Days 28 and 56 | 36 weeks
  Complete clinical remission with incomplete count recovery (CRi) at day 28 and 56 for study participants treated at the recommended phase 2 (RP2D) dose level, defined as complete clinical remission except with ANC< 1000/μL and/or platelets <100,000/μL
Complete Clinical Remission (CR) with Measurable Residual Disease (MRD) | 36 weeks
  Complete clinical remission with measurable residual disease (MRD) negativity at day 28 and 56 for participants treated at the recommended phase 2 (RP2D) dose level.
Complete clinical remission with incomplete count recovery (CRi) with Measurable Residual Disease (MRD) | 36 weeks
  CRi with MRD negativity at days 28 and 56, defined by absence of detectable disease by flow cytometry (sensitivity of 0.01%), and V(D)J next-generation sequencing-based MRD assessment (sensitivity of 0.0001%)
Overall Survival | 36 weeks
  Overall survival (OS), defined as the time from treatment administration to death from any cause, or until last contact if the patient has not died.
Progression-Free Survival | 36 weeks
  Progression-free survival (PFS), defined as the time from treatment administration to documented disease progression or death from any cause, or until last contact if no event has occurred.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF